CLINICAL TRIAL: NCT00559572
Title: Motivating Persons With Schizophrenia to Exercise
Brief Title: Effects of Motivating People With Schizophrenia to Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Brenda Lawson, Compliance Officer, IRB Administrator, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R03MH079047 (NIH); R03MH079047 (NIH)
Record Dates: First submitted 2007-11-14; First posted 2007-11-16 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Schizophrenia
Keywords: Exercise; Group Counseling; Obesity
MeSH Terms: conditions — Schizophrenia; Motor Activity; Obesity | interventions — Time

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Exercise information group
  Interventions: Behavioral: Motivational group sessions
- 2 (Active Comparator): General health information group
  Interventions: Other: Time and attention control group sessions

INTERVENTIONS:
Behavioral: Motivational group sessions — Motivational group sessions include 4 weeks of weekly 1-hour exercise information sessions.
  Arms: 1
Other: Time and attention control group sessions — Time and attention control group sessions include 4 weeks of weekly 1-hour general health information sessions.
  Arms: 2

SUMMARY:
This study will evaluate the impact of motivational guidance to exercise on people with schizophrenia, based on their participation in a walking program.

DETAILED DESCRIPTION:
Schizophrenia is a chronic brain disorder that affects about 1% of Americans. People with schizophrenia experience extreme paranoia, often claiming that they hear voices not heard by others and that others are invading or controlling their minds with the intent to hurt them. More specific symptoms include hallucinations, delusional behaviors, disordered movements, and decreased ability to comprehend and apply information to everyday activities. The severity of these symptoms makes self-care and regular exercise difficult for people with schizophrenia. The fatality rate from diabetes, heart disease, and other obesity-related illnesses is significantly higher in people with schizophrenia. Exercise is known to reduce health problems associated with obesity, yet few studies have encouraged exercise as a treatment method for improving the health of those with schizophrenia. Furthermore, the long-term physical and mental effects of consistent exercise on people with schizophrenia are not well-known. This study will evaluate the impact of motivational guidance to exercise on people with schizophrenia, based on their attendance, persistence, and compliance to a walking program.

Participants in this study will be randomly assigned to one of two groups. Both groups will continue their regular medications and treatments throughout the study. Upon entry, members of both groups will complete the same two forms concerning attitudes toward exercise. Group 1 participants will attend weekly 1-hour exercise information sessions for 4 weeks. Group 2 participants will attend weekly 1-hour general health information sessions for the same 4 weeks. Participants of both groups will then take part in identical 16-week walking programs. The walking program will consist of three 30- to 50-minute walks per week, including 10 minutes of warm up and 10 minutes of cool down stretching. All participants will gradually increase their walking time from 5 minutes to 30 minutes during the program. At the completion of the walking programs, participants of both groups will complete repeat forms about their attitudes toward exercise. There will be no follow-up visits for the participants.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for schizophrenia
* Speaks English
* Stable medication regimen
* Able to receive medical clearance for moderate exercise

Exclusion Criteria:

* Hospitalized within 1 year of study entry for angina, heart attack, or cardiac surgery
* Diagnosed with congestive heart failure
* Has a pacemaker
* Heart rate less than 50 bpm or more than 100 bpm at rest
* Uncontrolled hypertension
* History of spinal or hip fracture
* Unable to walk or move around without assistance
* Any other medical condition, in the opinion of primary care provider, that would prevent safe participation in the study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-11; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Exercise group attendance | Measured at Week 16
Exercise group persistence | Measured at Weeks 4,8, 12 & 16
Exercise group compliance | Measured at Weeks 4,8,12 & 16
Exercise attitude | Measured at Weeks 4,8,12 and 16

CONTACTS AND LOCATIONS:
Overall Officials: Lora L. Beebe, PhD, PMHNP, BC, Principal Investigator — University of Tennessee
Locations (1):
- Helen Ross McNabb Center, Knoxville, Tennessee, United States